CLINICAL TRIAL: NCT02727582
Title: Pharmacometric Optimization of Second Line Drugs for MDR Tuberculosis Treatment
Acronym: PODrtb
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Helen Margaret McIlleron, Senior Research Officer, University of Cape Town
Other Study IDs: PODrtb
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Multidrug-resistant Tuberculosis
Keywords: MDR
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multidrug-resistant (MDR) tuberculosis (TB), defined as simultaneous resistance to isoniazid and rifampin, has been declared a global emergency. Treatment outcomes are poor, driven by toxicity and limited efficacy of the 2nd-line anti-TB drugs.

Although there is evidence that both anti-TB activity and most of the toxicity of the key drugs are related to drug exposure, the pharmacokinetic/pharmacodynamic (PK/PD) relationships in patients with MDR-TB are poorly characterized. Moreover potential synergy of drug combinations has not been identified in the context of MDR-TB, dosing has not taken into account the concentrations needed to suppress resistance, and the role of minimum inhibitory concentrations (MICs) in dosing is poorly studied.

There are therefore opportunities to optimize drug doses and combinations to improve efficacy, and reduce toxicity. Based on this observational study of patients on standard treatment for MDR-TB, our proposal builds on novel methodologies we have developed, largely for drug sensitive TB:

1. The application of computational analytical techniques to tease out the individual contributions of anti-TB drugs used in combination
2. The development of a treatment response biomarker model based on time-to-positivity in liquid culture of serial sputum samples.
3. The in vitro determination of PK targets for anti-TB activity and the suppression of resistance using the hollow fiber models of Mycobacterium tuberculosis (Mtb) (HFM-TB).

Thus the research will enhance our understanding of current modalities of TB treatment, while contributing research approaches for future regimen optimization.

This protocol describes the clinical research component (points 1&2).

Aim 1: To characterize the effects of 2nd-line drug exposures on treatment response in MDR-TB patients. The 2nd-line drugs to be examined are those comprising the standardized regimen used in South Africa: kanamycin, pyrazinamide, moxifloxacin, ethionamide and terizidone.

Hypothesis: Amongst patients on standard MDR-TB treatment, variation in drug exposure has a quantifiable impact on the rates at which viable Mtb are cleared from the sputum.

Aim 2: To identify drug exposures associated with the risk of treatment-related toxicities in patients on a standard 2nd-line regimen for MDR-TB.

Hypothesis: The risks of specific toxicities associated with kanamycin, pyrazinamide, moxifloxacin, ethionamide and terizidone are linked to drug concentrations.

DETAILED DESCRIPTION:
Aim 1: To characterize the effects of 2nd-line drug exposures on treatment response in MDR-TB patients. The 2nd-line drugs to be examined are those comprising the standardized regimen used in South Africa: kanamycin, pyrazinamide, moxifloxacin, ethionamide and terizidone.

Hypothesis: Amongst patients on standard MDR-TB treatment, variation in drug exposure has a quantifiable impact on the rates at which viable Mtb are cleared from the sputum.

Rationale: There is substantial variability in the PK parameters of the 2nd-line drugs between patients, and in the susceptibility of individual Mtb isolates to those drugs. Concentration-dependent activity has been demonstrated for moxifloxacin, pyrazinamide and aminoglycosides, and higher doses of moxifloxacin and pyrazinamide have been proposed. Studies are needed to identify the most important determinants of treatment response and to describe the optimal drug exposures in MDR-TB, taking MICs into account. We will describe the exponential decline of viable Mtb in the sputum of MDR-TB patients in a treatment response model based on time-to-positivity in liquid culture, thus furthering the field of TB biomarker research. We will then define the relationship between PK and the rates of eradication of viable Mtb from the sputum of patients on the standard MDR-TB regimen to identify the more potent drugs driving treatment response, and to identify synergism or antagonism between individual drugs. Examples of specific questions that will be addressed include: What is the impact of pyrazinamide resistance on treatment response?; What is the impact of inhA mutations on the effect of ethionamide?; and, Should a higher doses of moxifloxacin and pyrazinamide be considered?

Aim 2: To identify drug exposures associated with the risk of treatment-related toxicities in patients on a standard 2nd-line regimen for MDR-TB.

Hypothesis: The risks of specific toxicities associated with kanamycin, pyrazinamide, moxifloxacin, ethionamide and terizidone are linked to drug concentrations.

Rationale: Treatment limiting adverse drug effects are common in patients on MDR-TB treatment regimens. Although several common toxicities are linked to specific drugs and are thought to be dose-related, the relationship between PK and toxicity has not been adequately studied. Overlapping toxicity of antiretroviral drugs in HIV-infected patients, amongst other risk factors, may be contributory. Minimum drug concentration thresholds associated with increased toxicity would allow optimization of doses by targeting concentrations below which toxicity is common, but above which there is optimal efficacy.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Current diagnosis of pulmonary MDR-TB or rifampicin-monoresistant TB

Baseline sputum sample with positive Gene Xpert MTB/RIF test, or confirmed positive Mycobacterium tuberculosis culture displaying resistance to rifampicin with or without isoniazid resistance on standard DST.

Eligible for standard MDR-TB treatment regimen (see Table 1), or, started on standard MDR-TB regimen within the past 1 month.

Written confirmation of informed consent to participate.

Pregnant women satisfying all other eligibility criteria may be enrolled.

Exclusion Criteria:

Critically ill or medically unstable* e.g. organ failure - on ventilator, receiving dialysis for acute renal failure, fulminant hepatitis (*can be recruited once stabilized if still eligible), or severe haemoptysis.

Unwilling to participate, or unable to understand the Participant information and provide full informed consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 142 Xpert MTB/RIF positive adults (>18 years of age), with or without HIV, and starting the standard 5-drug regimen for MDR-TB. The MDR-TB regimen also applies to patients who have rifampicin mono-resistant TB so these patients will also be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
To characterize the effects of 2nd-line drug exposures on treatment response in MDR-TB patients. | 2 years
  To describe the population PK of moxifloxacin, terizidone, ethionamide, pyrazinamide and kanamycin in a cohort of 142 South African patients diagnosed with MDR-TB.
  * Develop LC-MS/MS assays to accurately quantify moxifloxacin, terizidone, ethionamide, pyrazinamide and kanamycin in plasma.
  * Determine plasma concentrations of the 5 drugs in serial samples (6 samples drawn during a dosing interval) in each patient.
  * Develop population nonlinear mixed effects models to describe the plasma PK of the 5 drugs in patients with MDR-TB.
  * Estimate individual PK measures of exposure for each drug.
  * In those patients who consent to pharmacogenetic evaluation, collect and store a suitable blood sample

SECONDARY OUTCOMES:
To identify drug exposures associated with the risk of treatment-related toxicities in patients on a standard 2nd-line regimen for MDR-TB. | 2 years
  To describe the individual susceptibility and MIC distributions of the infecting strains of Mtb in the study population.
  • Determine moxifloxacin, kanamycin, ethionamide, isoniazid, cycloserine and pyrazinamide MICs in baseline culture isolates in each patient and in positive 8-week cultures

OTHER OUTCOMES:
Develop a treatment response model using time to positivity (TTP) in serial MGIT sputum cultures as a surrogate marker to quantify viable mycobacterial burden by time and hence response to treatment during the initial phase of treatment. | 2 years
  Using TTP data from serial MGIT cultures taken weekly during the first 12 weeks of treatment, to develop a nonlinear mixed effects model describing the population response to standard MDR-TB treatment.
  • Individual model parameter estimates will be obtained from the model
To describe the key drivers of treatment response in the standard multi-drug regimen for MDR-TB | 2 years
  * Quantify the effects of PK exposure and MIC on key treatment response parameters
  * Identify key PK thresholds for treatment response
Describe the safety and tolerability of standard MDR-TB treatment through serial standardized collection of laboratory results and AE data, and describe PK associations with such toxicity. | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Brooklyn Chest Hospital, Cape Town, Western Cape
  - DP Marias Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
The investigators listed on the protocol comprise the study management group and are the custodians of the data generated from the study. All manuscripts arising from the data generated as a result of this study are to be approved by this group before submission for publication. Manuscripts arising from the trial will be submitted to peer-reviewed journals. In accordance with NIH public access policy the final peer-reviewed journal manuscripts will be submitted NIH Manuscript Submission System (NIHMS) upon acceptance for publication, and be made publicly available on PubMed Central no later than 12 months after the official date of publication. All presentations and publications will acknowledge the trial's funding sources. Authorship will follow the recommendations of the International Committee of Medical Journal Editors (ICMJE) and the study management group will resolve any problems of authorship and maintain the quality of publications